CLINICAL TRIAL: NCT00838578
Title: Phase I/II Study of KRN330 Plus Irinotecan After First-Line or Adjuvant FOLFOX/CapOx Failure in Patients With Metastatic Colorectal Cancer
Brief Title: Phase I/II Study of KRN330 Plus Irinotecan in Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per protocol, the study was terminated based on interim analysis results
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRN330-US-02
Record Dates: First submitted 2009-02-04; First posted 2009-02-06 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
Keywords: KRN330; Colorectal Cancer; Antimetabolites; Antimetabolites, Antineoplastic; Digestive System Neoplasms; Immunologic Factors; Molecular Mechanisms of Pharmacological Action; Antineoplastic Agents; Gastrointestinal Diseases; Physiological Effects of Drugs; Colonic Diseases; Irinotecan; Enzyme Inhibitors; Intestinal Diseases; Immunosuppressive Agents; Rectal Diseases; Pharmacologic Actions; Intestinal Neoplasms; Neoplasms by Site; Digestive System Diseases; Therapeutic Uses; Fluorouracil; Neoplasms; Gastrointestinal Neoplasms; Antineoplastic Agents, Phytogenic; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms; Digestive System Neoplasms; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases; Intestinal Neoplasms; Neoplasms by Site; Digestive System Diseases; Neoplasms; Gastrointestinal Neoplasms | interventions — KRN-330; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KRN330 + Irinotecan (Experimental): open label, single arm
  Interventions: Biological: KRN330; Drug: Irinotecan

INTERVENTIONS:
Biological: KRN330 — KRN330 will be dosed at 0.5 mg/kg weekly until disease progression.
Drug: Irinotecan — Irinotecan will be dosed at 180 mg/m2 biweekly until disease progression.

SUMMARY:
The primary objective of the Phase II portion of this study is to assess the efficacy of KRN330 in combination with irinotecan after first-line or adjuvant FOLFOX (5-fluorouracil, leucovorin, and oxaliplatin)/CapOx (capecitabine and oxaliplatin) treatment failure in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
Phase II portion is an open-label, single arm study. Based on the results of the Phase I portion, weekly KRN330 (0.5 mg/kg) and biweekly irinotecan (180 mg/m2) will be used in the Phase II portion. To be eligible for the Phase II portion, a patient will have recurred or progressed within 6 months of the last cycle of FOLFOX/CapOx +/- bevacizumab (first-line or adjuvant regimen for metastatic colorectal cancer). Patients will continue the treatment until disease progression.

Per protocol, the decision was made to terminate the study based on interim analysis results. The Response Rate in Phase II did not meet the protocol-specified RR of 15% when 0.5 mg/kg KRN330 was administered weekly in combination with irinotecan(180 mg/m2)biweekly.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed colorectal cancer that is metastatic with measurable disease.
* For the Phase II portion: Have recurred or progressed within 6 months of the last cycle of FOLFOX +/- bevacizumab first-line or adjuvant regimen for metastatic colorectal cancer. Note: Those who had initiated FOLFOX/CapOx but stopped oxaliplatin because of intolerable toxicity are also eligible.
* At least 4 weeks have elapsed since the last chemotherapy, radiotherapy, immunotherapy, or biologic therapy prior to enrollment (except at least 6 weeks in the case of nitrosourea and mitomycin).
* Have not received any other investigational agents within 4 weeks of study entry and have fully recovered from any adverse event due to prior therapy.
* At least 4 weeks have elapsed since any major surgery.
* Have ECOG performance status of 0, 1, or 2.
* Have adequate bone marrow and organ function

Exclusion Criteria:

* Have an active, uncontrolled infection.
* Have known HIV positive status.
* Have known or suspected cerebral metastasis.
* Have had a myocardial infarction (MI) or cerebrovascular accident (CVA) within the last 6 months; or meet the criteria for AHA class III or IV congestive heart failure (CHF).
* Have a medical condition requiring chronic use of high-dose corticosteroids or other chronic immunosuppressive therapy (e.g. methotrexate, azathioprine).
* Have a history of greater than or equal to Grade 2 allergic reaction or hypersensitivity following exposure to humanized or human monoclonal antibodies (but not chimeric antibodies).
* Pregnant or breastfeeding women and male or female patients who do not agree to use effective contraceptive method(s) during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-03; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kurman, MD, Study Director — Kyowa Hakko Kirin Pharma, Inc.
Locations (12):
- United States (12):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Arizona Clinical Research Center, Tucson, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Lombardi Comprehensive Cancer Center, Georgetown University Hospital, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Fort Myers, Florida
  - University of Florida COllege of Medicine/Shands Cancer Center, Gainesville, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - NYU Clinical Trials Office, New York University Cancer Institute, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- KRN330 + Irinotecan: * Phase 1____ Biweekly KRN330 (0.5 mg/kg) (N=8) Weekly KRN330 (0.5 mg/kg) (N=7) Biweekly KRN330 (1.0 mg/kg) (N=4) Total (N=19)
  * Phase 2____ Weekly KRN330 (0.5 mg/kg)) (N=46)
  Phase 1 and 2Combined (N=65)
Period: Overall Study
Arm/Group | KRN330 + Irinotecan
Started | 65 (In this Ph 1/2 study, 65 subjects were enrolled; 2 were protocol violators, so only 63 treated.)
Completed | 63
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | KRN330 + Irinotecan
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.83 (10.185)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious and Other (Non-Serious) Adverse Events According to the CTCAE v.3.0
Time Frame: Until disease progression, death, or withdrawal post initial KRN330 treatment, assessed up to 100 months
Population: ITT population
Measure: Number; unit: participants
Groups:
- Regimen A: KRN330 Biweekly + Irinotecan Biweekly: In treatment regimen A, both KRN330 and irinotecan (180 mg/m2) were administered biweekly(Weeks 1, 3, and 5).
  Cohort 1: 1 mg/kg KRN330 biweekly and 180 mg/m2 irinotecan biweekly Cohort 2: 0.5 mg/kg KRN330 biweekly and 180 mg/m2 irinotecan biweekly
- Regimen B: KRN330 Weekly + Irinotecan Biweekly: treatment regimen B, KRN330 was administered weekly (Weeks 1, 2, 3, 4 and 5) and irinotecan (180 mg/m2) biweekly (Weeks 1, 3, and 5).
- PH 2 Treatment: KRN330 Wkly + IRI Biwkly: The Phase 2 portion was a single arm study using the regimen and dose selected in Phase 1 (0.5 mg/kg KRN330 weekly and 180 mg/m2 irinotecan biweekly).
Arm/Group | Regimen A: KRN330 Biweekly + Irinotecan Biweekly | Regimen B: KRN330 Weekly + Irinotecan Biweekly | PH 2 Treatment: KRN330 Wkly + IRI Biwkly
Number analyzed (Participants) | 12 | 7 | 44
participants | 12 | 7 | 44

ADVERSE EVENTS:
Groups:
- Phase 1 Regimen A: KRN330 Biweekly + IRI Biweekly: In Regimen A, patients received both KRN330 and irinotecan biweekly (Weeks 1, 3, and 5):
  Cohort 1: KRN330 1.0 mg/kg + irinotecan 180 mg/m2 Cohort 2: KRN330 0.5 mg/kg + irinotecan 180 mg/m2
- Phase 1 Regimen B: KRN330 Weekly + IRI Biweekly: In Regimen B, patients received KRN330 0.5 mg/kg weekly (Weeks 1, 2, 3, 4, and 5) and irinotecan 180 mg/m2 biweekly (Weeks 1, 3, and 5)
- Phase 2: KRN330 Weekly + IRI Biweekly: The Phase 2 portion had a single arm in which patients received Regimen B as included in the Phase 1 portion
Arm/Group | Phase 1 Regimen A: KRN330 Biweekly + IRI Biweekly | Phase 1 Regimen B: KRN330 Weekly + IRI Biweekly | Phase 2: KRN330 Weekly + IRI Biweekly
Serious Adverse Events (participants affected / at risk) | 6/12 | 2/7 | 17/44
Other Adverse Events (participants affected / at risk) | 12/12 | 7/7 | 42/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Regimen A: KRN330 Biweekly + IRI Biweekly (N=12) | Phase 1 Regimen B: KRN330 Weekly + IRI Biweekly (N=7) | Phase 2: KRN330 Weekly + IRI Biweekly (N=44)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 4 (4)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2)
Disease progression (General disorders) | 0 (0) | 0 (0) | 8 (8)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile toxin test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metastatic pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Regimen A: KRN330 Biweekly + IRI Biweekly (N=12) | Phase 1 Regimen B: KRN330 Weekly + IRI Biweekly (N=7) | Phase 2: KRN330 Weekly + IRI Biweekly (N=44)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (2) | 10 (16)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 8 (16)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 7 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 7 (7)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Swollen tear duct (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (7) | 3 (7) | 14 (22)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Abdominal wall mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4) | 1 (3) | 13 (24)
Diarrhoea (Gastrointestinal disorders) | 10 (17) | 5 (12) | 33 (73)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (13) | 6 (17) | 29 (55)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Rectal discharge (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 5 (9) | 6 (12) | 17 (28)
Application site rash (General disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 5 (7)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 2 (3)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (5) | 4 (11) | 29 (54)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 2 (2)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 9 (13)
Pain (General disorders) | 0 (0) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 7 (7)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 2 (4)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Lice infestation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 1 (1) | 6 (6)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Procedural site reaction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 5 (5)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 2 (3) | 0 (0) | 1 (2)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 3 (4)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 2 (2)
Clostridium difficile toxin test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 3 (6)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Skin turgor decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 2 (3) | 5 (9)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 2 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 15 (25)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 14 (27)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 3 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 5 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cholinergic syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 8 (11)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 4 (6)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (4)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 5 (6)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (4)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (4) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Scrotal erythema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (5) | 7 (8)
Dysphonia (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 7 (8)
Epistaxis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Rhinorrhoea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 17 (20)
Dandruff (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 4 (9)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (6) | 8 (22)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 6 (6)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other